CLINICAL TRIAL: NCT00251394
Title: A Phase 2, Open-Label Study of the Efficacy, Safety, and Tolerability of Dynavax's Immunostimulatory Phosphorothiolate Oligodeoxyribonucleotide, 1018 ISS, Following Rituxan (Rituximab) Treatment in Patients With CD20+, B-Cell Follicular Non-Hodgkin's Lymphoma.
Brief Title: Study of Dynavax's 1018 ISS, Following Rituxan in Patients With B-Cell Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Dynavax Technologies Corporation (Industry); James P. Wilmot Cancer Center (Other); University of Rochester (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Arnold Freedman, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-411; R21; U10402
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2009-07

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: B-Cell follicular non-Hodgkin's lymphoma; Rituxan; Rituximab; 1018 ISS; CD 20 +
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; 1018 oligonucleotide

INTERVENTIONS:
Drug: Rituxan — Given intravenously once weekly for four weeks.
Drug: 1018 ISS — Given as an injection under the skin after the 2nd, 3rd and 4th rituxan infusion. One week after the last rituxan infusion is given, a fourth and final 1018ISS injection will be given.

SUMMARY:
The main purpose of this study is to determine the effects (good and bad) and the safety of Dynavax's immunostimulatory phosphorothiolate oligodeoxyribonucleotide (1018 ISS) given in combination with Rituxan on patients with B-cell follicular non-Hodgkin's lymphoma. This research is being done because recurrent follicular non-Hodgkin's lymphoma is not curable with standard chemotherapy or antibody treatments. 1018 ISS is an experimental compound that consists of short pieces of DNA that stimulate the immune system. It is hoped that 1018 ISS may improve the ability of Rituxan to kill cancer cells.

DETAILED DESCRIPTION:
* Patients will receive four weekly infusions of Rituxan which is standard treatment for B-cell non-Hodgkin's lymphoma. Approximately 30 to 60 minutes after the second, third and fourth infusions of Rituxan, the patient will receive up to 3 injections of 1018 ISS under the skin. The number of injections will depend upon the patients weight. One week after the last Rituxan infusion the patient will receive a fourth and final injection of 1018 ISS.
* After completion of the 5-week treatment period, a physical examination and blood work will be performed. The patient will also be examined to see if the tumor has gotten smaller, bigger, or stayed the same size and in the same places by either CT scan or MRI. A bone marrow aspiration and biopsy will be done to examine any changes in bone marrow cells.
* The following tests will be performed to determine whether or not a patient is eligible to participate in this clinical study: Bone marrow aspiration and biopsy; lymph node biopsy; skin biopsy; standard x-ray tests (x-rays, CT scans, MRI, ultrasounds, and/or radioactive drug scans); and blood work.
* While receiving treatment patients will have the following procedures done; Physical examination once a week for 4 weeks, blood testing for any changes in the blood, blood chemistry and other blood components. Patients will also be requested to keep a diary between each study visit to record any health changes or any over-the-counter medication or herbal preparation they may have taken.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Pathological evidence of CD20+, B-cell follicular non-Hodgkin's lymphoma
* Received at least one previous chemotherapy regimen for lymphoma
* Hemoglobin > 8.5 g/dl
* WBC > 2,000/mm3
* ANC > 1,000/mm3
* Platelet count > 75,000/mm3
* ECOG performance status of less than or equal to 2
* Life expectancy of greater than 4 months
* Women and men of childbearing potential must be willing to use highly effective methods of birth control for duration of time on the study

Exclusion Criteria:

* Pregnant of lactating women
* Treatment with chemotherapy, including systemic steroids, or radiation therapy within 30 days
* Current use of systemic or inhaled steroids
* Treatment with radioimmunotherapy, autologous stem cell transplantation, or fludarabine within 6 months
* Disease progression within 6 months of any previous rituximab therapy
* History of allogenic transplantation, including nonmyeloablative transplantation
* Unstable angina, symptomatic cardiac arrhythmia or clinical heart failure
* Severe pulmonary disease, symptomatic pleural effusions, or clinically significant pulmonary symptoms
* Active infection requiring systemic antibiotic, antiviral, or antifungal therapy
* Clinically apparent CNS lymphoma
* Major surgery within 2 weeks
* Known human anti-murine antibody (HAMA) or human anti-chimeric antibody (HACA) response
* Known Hepatitis B surface antigen positive
* History of autoimmune disorder
* Current therapeutic use of anticoagulants
* History of coagulopathy
* Known allergy to any of the components of 1018 ISS or Rituxan
* Participation in another investigational trial within 30 days
* Any clinically significant abnormality in screening blood chemistry, hematology, or urinalysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2006-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of patients who are alive and without disease progression 1 year after initiating Rituxan plus 1018 ISS therapy. | 2 years

SECONDARY OUTCOMES:
To assess the overall response rate following treatment | 2 years
to determine duration of response and time to progression
to further define the safety profile of 1018 ISS | 2 years
to explore the biologic activity of 1018 ISS. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Freedman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts